CLINICAL TRIAL: NCT00365482
Title: Bipolar Disorder in Epilepsy
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 06.02.029
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsy; Bipolar Disorder
Keywords: Epilepsy; Bipolar Disorder
MeSH Terms: conditions — Epilepsy; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out how often major mood swings occur in patients treated in a specialty epilepsy center.

DETAILED DESCRIPTION:
Bipolar disorder (a condition of major mood swings) or milder forms of ups and downs in mood may occur with a number to neurological conditions. Recently, one study showed that these mood changes occur fairly often in individuals with epilepsy studied in the general community. We speculate that bipolar symptoms occur with even higher frequency in a tertiary epilepsy center than that encountered in the previous community-based study. The goals of this study are to assess:

* the rate of bipolar symptoms as measured by a self-reporting screening tool in a tertiary epilepsy center setting
* the meaning of a positive screening score in epilepsy patients
* the utility, sensitivity and specificity of alternative screening tools for mood instability in epilepsy patients
* the correlation of mood instability with seizure-related variables
* the relation of a positive screening score on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Being evaluated at the Long Island Jewish Comprehensive Epilepsy Center
* Capable of completing self-reporting questionnaires

Exclusion Criteria:

* Patients with mental retardation
* Patients with pseudoseizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Epilepsy patients at the Long Island Jewish Comprehensive Epilepsy Center
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Hwang, MD, Principal Investigator — Long Island Jewish Medical Center
Locations (1):
- North Shore Long Island Jewish Health System, Great Neck, New York, United States